CLINICAL TRIAL: NCT03927105
Title: Nivolumab and the Antagonistic CSF-1R Monoclonal Antibody Cabiralizumab (BMS-986227) in Patients With Relapsed/Refractory Peripheral T Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-HEM16-085
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2021-09-10 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Nivolumab; cabiralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Cabiralizumab (Experimental): Nivolumab 240mg IV + Cabiralizumab 4mg/kg on day 1 of every 14 day cycle.
  Interventions: Drug: Nivolumab; Drug: cabiralizumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a human monoclonal antibody (HuMAb; immunoglobulin G4 [IgG4]-S228P) that targets the programmed death-1 (PD-1) cluster of differentiation 279 (CD279) cell surface membrane receptor. PD-1 is a negative regulatory molecule expressed by activated T and B lymphocytes.1 Binding of PD-1 to its ligands, programmed death-ligands 1 (PD-L1) and 2 (PD-L2), results in the down-regulation of lymphocyte activation. Inhibition of the interaction between PD-1 and its ligands promotes immune responses and antigen-specific T-cell responses to both foreign antigens as well as self-antigens. Nivolumab will be delivered intravenously at a fixed dose of 240 mg on day 1 of 14 day cycles.
  Other Names: Opdivo; BMS-936558; MDX1106
Drug: cabiralizumab — Cabiralizumab is a recombinant, humanized Immunoglobulin G4 (IgG4) monoclonal antibody that binds to human colony stimulating factor 1 receptor (CSF1R; c-fms). Cabiralizumab will be delivered intravenously at a dosage of 4 mg/kg on day 1 of 14 day cycles.
  Other Names: BMS-986227; FPA008

SUMMARY:
A multicenter trial evaluating the combination of nivolumab and the antagonistic CSF-1R monoclonal antibody cabiralizumab (BMS-986227) in patients with relapsed/refractory peripheral T cell lymphoma

DETAILED DESCRIPTION:
Enrollment to this study was discontinued after four subjects due to industry-related changes to the Cabiralizumab program.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for clinical trial enrollment and mandatory consent for any biopsies as well as HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-2.
* Histological confirmation of peripheral T-cell lymphoma (PTCL) except adult T-cell leukemia/lymphoma (ATLL).
* Documented disease progression after receiving at least two prior therapeutic regimen including brentuximab vedotin in patients with CD30 positive disease (defined as >10% CD30 positive cells).
* Prior cancer treatment must be completed at least 28 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤ grade 1 or baseline. Systemic steroids at a dose less than the equivalent of 10 mg/day of prednisone and inhaled, nasal, and topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease are permitted. Treatment with a short course of steroids (< 5 days) up to 7 days prior to study registration is permitted. Intermittent dexamethasone for the treatment of nausea/emesis is also permitted.
* Demonstrate adequate organ function as defined in the table in the protocol; all screening labs to be obtained within 28 days prior to registration.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L or equivalent units of human chorionic gonadotropin) performed at screening and within 24 hours of first dose of investigational treatment. See Section 5.4.1 of the protocol for definition of childbearing potential.
* Females of childbearing potential must be willing to abstain from heterosexual activity or use an effective method of contraception from the time of informed consent until 5 months after the last dose of investigational product. See Section 5.4.1 of the protocol for methods of contraception.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving study drugs and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. See Section 5.4.1 of the protocol for methods of contraception.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* PTCL histology consistent with ATLL.
* A history of, or a concurrent, clinically significant illness, medical condition or laboratory abnormality that, in the investigator's opinion, could affect the conduct of the study.
* Active infection requiring systemic therapy
* Recent (<100 days) autologous stem cell transplant, or previous allogeneic stem cell transplant.
* Known positive test for HIV. NOTE: HIV screening is not required.
* History of any chronic hepatitis as evidenced by the following:

  * Positive test for hepatitis B surface antigen
  * Positive test for qualitative hepatitis C viral load (by polymerase chain reaction [PCR]).
  * NOTE: Participants with positive hepatitis C antibody and negative quantitative hepatitis C by PCR are eligible. History of resolved hepatitis A virus infection is not an exclusion criterion.
* Pregnant or breastfeeding. NOTE: breast milk cannot be stored for future use while the mother is being treated on study.
* Previous malignancies (except non-melanoma skin cancers and in situ bladder, gastric, colorectal, endometrial, cervical/dysplasia, melanoma, or breast cancers) unless complete remission was achieved at least 2 years prior to study entry and no additional therapy is required during the study period.
* Prior treatment with cabiralizumab (or other CSF1R pathway inhibitors).
* Prior treatment with nivolumab or other medications within the checkpoint blockade family.
* Any unregulated nutritional or herbal supplement or recreational drug within 2 weeks prior to registration which, in the opinion of the study investigator, has the potential to cause hepatic injury.
* Concomitant use of statins for treatment of hypercholesterolemia. Statins are allowed only if the patient is on a stable dose for over 3 months prior to study registration and is in a stable status without CK elevations.
* Non-oncology vaccine therapies for prevention of infectious diseases (e.g., human papilloma virus vaccine) within 4 weeks of study registration. The inactivated seasonal influenza vaccine can be given to patients before treatment and while on therapy without restriction. Influenza vaccines containing live virus or other clinically indicated vaccinations for infectious diseases (i.e., pneumovax, varicella, etc.) may be permitted, but must be discussed with the sponsor investigator and may require a study drug washout period before and after administration of vaccine.
* Known history of sensitivity to infusions containing Tween 20 (polysorbate 20) and Tween 80 (polysorbate 80)
* History of allergy to any components of cabiralizumab or nivolumab
* Active, known, or suspected autoimmune disease.

  * NOTE: Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study treatment), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll after discussing with the sponsor investigator.
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity.
* Current or history of clinically significant muscle disorders (e.g., myositis), recent unresolved muscle injury, or any condition known to elevate serum CK levels.
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction or stroke/transient ischemic attack within the past 6 months
  * Uncontrolled angina within the past 3 months
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  * History of other clinically significant heart disease (e.g., cardiomyopathy (impaired LVEF), congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, significant pericardial effusion, or myocarditis)
  * Cardiovascular disease-related requirement for daily supplemental oxygen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Wilcox, MD, PhD, Principal Investigator — University of Michigal Rogel Cancer Center
Locations (3):
- United States (3):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Unviersity of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant consented, was deemed eligible, and enrolled to the trial, however subject was never treated due to new medical problems causing ineligibility prior to treatment.
Groups:
- Nivolumab + Cabiralizumab: Nivolumab is a human monoclonal antibody (HuMAb; immunoglobulin G4 [IgG4]-S228P) that targets the programmed death-1 (PD-1) cluster of differentiation 279 (CD279) cell surface membrane receptor. PD-1 is a negative regulatory molecule expressed by activated T and B lymphocytes.1 Binding of PD-1 to its ligands, programmed death-ligands 1 (PD-L1) and 2 (PD-L2), results in the down-regulation of lymphocyte activation. Inhibition of the interaction between PD-1 and its ligands promotes immune responses and antigen-specific T-cell responses to both foreign antigens as well as self-antigens. Nivolumab will be delivered intravenously at a fixed dose of 240 mg on day 1 of 14 day cycles.
  Cabiralizumab is a recombinant, humanized Immunoglobulin G4 (IgG4) monoclonal antibody that binds to human colony stimulating factor 1 receptor (CSF1R; c-fms). Cabiralizumab will be delivered intravenously at a dosage of 4 mg/kg on day 1 of 14 day cycles.
Period: Overall Study
Arm/Group | Nivolumab + Cabiralizumab
Started | 4
Began Treatment | 3
Follow-up | 3
Completed (completed through primary outcome measure collection; two participants are still in observation for secondary outcome measure assessments (not yet completed).) | 0
Not Completed | 4
Not completed — Death | 1
Not completed — In observation for potential re-treatment | 2
Not completed — Subject was never treated due to new medical problems causing ineligibility prior to treatment. | 1

BASELINE CHARACTERISTICS:
Population: All subject consented, confirmed to be eligible, and registered to the trial.
Groups:
- Nivolumab + Cabiralizumab: Nivolumab 240mg IV + Cabiralizumab 4mg/kg on day 1 of every 14 day cycle.
  Nivolumab is a human monoclonal antibody (HuMAb; immunoglobulin G4 [IgG4]-S228P) that targets the programmed death-1 (PD-1) cluster of differentiation 279 (CD279) cell surface membrane receptor. PD-1 is a negative regulatory molecule expressed by activated T and B lymphocytes.1 Binding of PD-1 to its ligands, programmed death-ligands 1 (PD-L1) and 2 (PD-L2), results in the down-regulation of lymphocyte activation. Inhibition of the interaction between PD-1 and its ligands promotes immune responses and antigen-specific T-cell responses to both foreign antigens as well as self-antigens.
  Cabiralizumab is a recombinant, humanized Immunoglobulin G4 (IgG4) monoclonal antibody that binds to human colony stimulating factor 1 receptor (CSF1R; c-fms).
Arm/Group | Nivolumab + Cabiralizumab
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 62.5 [49 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at Four Months (LYRIC Criteria)
Description: Overall Response Rate (CR + PR) as determined by LYRIC (LYmphoma Response to Immunomodulatory therapy Criteria), at four months (shown as number of participants with CR or PR at 4 months).
  LYRIC: An adaptation of the Lugano classification developed because discriminating true progressive disease from pseudoprogression in lymphoma patients receiving immunomodulatory agents is challenging. To address this challenge, the LYRIC criteria incorporated the response category of "indeterminate response" (IR).
  * IR(1): ≥ 50% increase in overall tumor burden (sum of the product of the perpendicular diameters (SPD) of up to 6 target measurable nodes and extranodal sites) occurred in the 1st 12 weeks of therapy and without clinical deterioration
  * IR(2): new lesions or ≥ 50% increase of existing lesion(s) without a ≥ 50% increase of overall tumor burden at any time during treatment.
  * IR(3): increased FDG uptake of 1or more lesions without any increase in size or number of those lesions.
Time Frame: 4 months
Population: All subjects with measurable disease who received at least one cycle of treatment and had disease re-evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabiralizumab
Number analyzed (Participants) | 3
Participants
  Complete Response | 2
  Partial Response | 0
  Non-Responder | 1

2. Primary Outcome: Complete Response Rate (CRR) at Four Months
Description: Complete response rate, as determined by LYRIC criteria, at four months (reported as number of participants with CR at 4 months).
  LYRIC: An adaptation of the Lugano classification developed because discriminating true progressive disease from pseudoprogression in lymphoma patients receiving immunomodulatory agents is challenging. To address this challenge, the LYRIC criteria incorporated the response category of "indeterminate response" (IR).
  * IR(1): ≥ 50% increase in overall tumor burden (sum of the product of the perpendicular diameters (SPD) of up to 6 target measurable nodes and extranodal sites) occurred in the 1st 12 weeks of therapy and without clinical deterioration
  * IR(2): new lesions or ≥ 50% increase of existing lesion(s) without a ≥ 50% increase of overall tumor burden at any time during treatment.
  * IR(3): increased FDG uptake of 1or more lesions without any increase in size or number of those lesions.
Time Frame: 4 months
Population: All subjects with measurable disease who received at least one cycle of treatment and had disease re-evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabiralizumab
Number analyzed (Participants) | 3
Participants | 2

3. Secondary Outcome: Overall Response at Four Months by (LUGANO 2014) Criteria
Description: Overall response (CR + PR), as determined by LUGANO 2014 criteria (reported as number of participants with a CR or PR at 4 months).
  The Lugano classification is utilized for both lymphoma staging and response assessment and incorporates PET-CT imaging. Responses are described as either partial or complete, with a complete response requiring disappearance of metabolically active sites of disease.
Time Frame: four months
Population: All subjects with measurable disease who received at least one cycle of treatment and had disease re-evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabiralizumab
Number analyzed (Participants) | 3
Participants
  Complete Response | 2
  Partial Response | 0
  Non-Responder | 1

4. Secondary Outcome: Complete Response Rate at Four Months (LUGANO 2014) Criteria
Description: Complete Response Rate, as determined by LUGANO 2014 criteria, at (reported as number of participants with a CR at 4 months).
  The Lugano classification is utilized for both lymphoma staging and response assessment and incorporates PET-CT imaging. A complete response requires disappearance of metabolically active sites of disease.
Time Frame: four months
Population: All subjects with measurable disease who received at least one cycle of treatment and had disease re-evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabiralizumab
Number analyzed (Participants) | 3
Participants | 2

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival will be measured from date of enrollment until the criteria for disease progression (PD) is met or death occurs. Subjects who have not progressed will be right-censored at the date of the last disease evaluation.
Time Frame: Up to one year post treatment discontinuation or an estimated maximum of 60 months
Reporting Status: Not Posted

6. Secondary Outcome: Disease Control Rate (DCR)
Description: The proportion of all subjects with stable disease (SD) for 8 weeks, PR, or CR.
Time Frame: Up to one year post treatment discontinuation or an estimated maximum of 60 months
Reporting Status: Not Posted

7. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response measured from the time that measurement criteria are met for CR or PR (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since treatment started).
Time Frame: Up to one year post treatment discontinuation or an estimated maximum of 60 months
Reporting Status: Not Posted

8. Secondary Outcome: Time to Next Treatment (TNT)
Description: Time to next treatment (TNT) is defined as the time from the date of enrollment to the institution of next treatment.
Time Frame: Up to one year post treatment discontinuation or an estimated maximum of 60 months
Reporting Status: Not Posted

9. Secondary Outcome: Summarize Adverse Events
Description: Assess and summarize adverse events (AEs) using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: Up to 100 days post treatment discontinuation or an estimated maximum of 60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From time of consent through 100 days post treatment discontinuation. Longest actual collection for AEs: 13 months
Description: An AE is any untoward medical occurrence whether or not related to the study drug that appears to change in intensity during the course of the study.
  Abnormal laboratory values or diagnostic test results constitute AEs only if they induce clinical signs or symptoms or require treatment or further diagnostic tests Hospitalization for elective surgery or routine clinical procedures that are not the result of an AE (e.g.,surgical insertion of central line) should not be recorded as an AE.
Arm/Group | Nivolumab + Cabiralizumab
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab + Cabiralizumab (N=3)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
ENDOCARDITIS INFECTIVE (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab + Cabiralizumab (N=3)
PERIORBITAL EDEMA (Eye disorders) | 2 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (4)
NAUSEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHILLS (General disorders) | 1 (1)
FATIGUE (General disorders) | 2 (2)
FEVER (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (2)
WEIGHT LOSS (Investigations) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 2 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Liposarcoma
HEADACHE (Nervous system disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03927105/Prot_SAP_000.pdf